CLINICAL TRIAL: NCT06645665
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of Respiratory Syncytial Virus IN006 Bivalent mRNA Vaccine (IN006) in Healthy Adult Aged 18 Years and Above
Brief Title: A Study to Describe the Safety and Immunogenicity of a Respiratory Syncytial Virus Vaccine IN006 in Healthy Adult Aged 18 Years and Above
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Shenxin Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IN006002
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: mRNA Vaccine; IN006; Respiratory syncytial virus; Viral Diseases; Messenger RNA; Innorna; Shenxin; Vaccines; Respiratory tract infections; Safety; Reactogenicity; Immunogenicity; RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Virus Diseases; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Dose A in Younger Adults (Experimental): Single injection of Dose A of IN006 or matching-placebo on Day 0
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 2: Dose B in Younger Adults (Experimental): Single injection of Dose B of IN006 or matching-placebo on Day 0.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 3: Dose C in Younger Adults (Experimental): Single injection of Dose C of IN006 or matching-placebo on Day 0.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 4: Dose A in Older Adults (Experimental): One injection of either Dose A of IN006 or matching-placebo on Day 0. Participants who initially assigned to receive IN006 on Day 0 will be further randomized to receive a second injection of either IN006 or matching-placebo approximately 12 months later.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 5: Dose B in Older Adults (Experimental): One injection of either Dose B of IN006 or matching-placebo on Day 0. Participants who initially assigned to receive IN006 on Day 0 will be further randomized to receive a second injection of either IN006 or matching-placebo approximately 12 months later.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 6: Dose C in Older Adults (Experimental): One injection of either Dose C of IN006 or matching-placebo on Day 0. Participants who initially assigned to receive IN006 on Day 0 will be further randomized to receive a second injection of either IN006 or matching-placebo approximately 12 months later.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo

INTERVENTIONS:
Biological: Bivalent RSV Vaccine (IN006) — Formulation for injection
Biological: Placebo — 0.9% sodium chloride (normal saline) injection

SUMMARY:
The study will evaluate the safety, tolerability, and immunogenicity of 3 dose levels of IN006 in healthy adults aged 18 Years and Above; of a revaccination of IN006 given approximately 12 months after the initial vaccination in older adults (aged ≥60 years).

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy people aged 18-59 (Part 1) or ≥60 (Part 2), male or female.
2. Body mass index (BMI) in the range of 18 to 29 kg/m^2.
3. Laboratory tests, 12-lead electrocardiogram, chest radiograph, vital signs and physical examination results are normal during the screening period, or abnormal results assessed by the investigator had no clinical significance; Subjects ≥60 years old with stable medical conditions, whose risk was considered controllable by the investigator, could also be enrolled.
4. Women of childbearing age took effective contraception within 2 weeks before joining the study, and the pregnancy test results before vaccination are negative. All male and female subjects of reproductive age voluntarily agree to use effective contraception from the signing of informed consent until 6 months after vaccination.

Key Exclusion Criteria:

1. The results of vital signs show: for subjects with no history of hypertension or hypotension, systolic blood pressure ≥140mmHg or < 90mmHg, and/or diastolic blood pressure ≥90mmHg or < 50mmHg; for subject with a history of hypertension not appropriately controlled via pharmaceutical treatment, systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg in those aged 40-59, and systolic blood pressure ≥150mmHg or diastolic blood pressure ≥90mmHg in those aged 60 and above. Pulse rate > 100 beats/min or < 50 beats/min; Ear temperature/oral temperature > 37.5°C (or axillary temperature > 37.0°C).
2. Laboratory tests, 12-lead electrocardiogram, chest radiography (orthographic) and physical examination results: For subjects aged 18-59 years old, abnormal results judged to be clinically significant by the investigator, or for subjects ≥60 years old, abnormal results judged to be > Grade 1 criteria by the investigator; For laboratory tests, a retest may be conducted at the discretion of investigators to determine subjects eligibility.
3. Those with tattoos, scars and ecchymosis at the injection site.
4. Known allergy to the experimental vaccine or its excipient, or history of severe allergy to other vaccines, foods, drugs, etc.
5. The subject has received any previous investigational or marketed RSV vaccine, or has received investigational or marketed RSV prophylactic monoclonal antibody within the last 6 months.
6. Received inactivated, subunit, or recombinant influenza vaccine within 14 days prior to enrollment, or received any live vaccine, nucleic acid vaccine, or adenovirus vector vaccine within 28 days prior to enrollment; Or plan to receive other vaccines within 28 days of vaccination.
7. Used antipyretic, analgesic or anti-allergic drugs within 3 days before enrollment.
8. Have received blood or blood-related products (including immunoglobulins) within 3 months prior to enrollment, or had planned to use them during the study period.
9. People with the following diseases:

   * A history of acute respiratory infection within 2 weeks of vaccination or a history of confirmed RSV-associated respiratory infection within 3 months prior to vaccination;
   * History of congenital or acquired immune deficiency or autoimmune disease, or long-term use (continuous use > 14 days) of corticosteroids (dose ≥20mg/ day prednisone or equivalent dose) or other immunosuppressants within the past 6 months;
   * people who are known to have been diagnosed with or currently have infectious diseases (including hepatitis B, hepatitis C, syphilis, and acquired immunodeficiency syndrome), or whose test positive for any of the hepatitis B surface antigens, hepatitis C antibodies, treponema pallidum antibodies, or human immunodeficiency virus antibodies;
   * A history or family history of neurological disease (convulsions, seizures, etc.); History or family history of mental illness;
   * Asplenia, or functional asplenia;
   * A history of myocarditis, pericarditis, or idiopathic cardiomyopathy, or any condition that increases the risk of myocarditis or pericarditis;
   * History of inflammatory demyelinating neuropathy such as Guillain-Barre syndrome;
   * Severe cardiovascular diseases, diabetes, blood and lymphatic system diseases, immune system diseases, liver and kidney diseases, respiratory diseases, metabolic and skeletal diseases, or malignant tumors (excluding stable chronic medical history, such as diabetes, hypertension, etc.);
   * Contraindications to intramuscular injection and blood drawing;
   * A history of tuberculosis (TB) or a positive T-cell test for TB infection (T-SPOT).
10. Had a history of major surgery within 3 months prior to vaccination or planned surgery during the trial.
11. Abuser of Drug or alcohol in the year prior to screening, which the investigator believes that it may impact on subjects' safety assessment or compliance.
12. Women of childbearing age who are breastfeeding, pregnant, have positive pregnancy test results or plan to become pregnant within 6 months after participating in the study.
13. Those who have received a vaccine or drug involving lipid nanoparticles (LNP) within 1 year, are participating in other RSV-related clinical trials, and are in or plan to participate in other clinical trials during the study period.
14. The investigator assesses that the subject has any disease or condition that would place the subject at an unacceptable risk; The subject is unable to meet protocol requirements; Conditions that interfere with the assessment of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Solicited Local and Systemic Adverse Reactions Through 14 Days After Initial Vaccination | From initial vaccination up to14 days post initial vaccination
Percentage of Participants With Unsolicited Adverse Events (AEs) Through 28 Days After Initial Vaccination | From initial vaccination up to 28 days post initial vaccination
Percentage of Participants With AEs Through 30 Minutes After Initial Vaccination | From initial vaccination up to 30 minutes post initial vaccination
Percentage of Participants With Any Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) During Study | Through study completion, about 2 years at most
Percentage of Abnormal Results of Hematology On Day 3 After Initial Vaccination Compared with Baseline | From initial vaccination up to day 3 post initial vaccination
Percentage of Abnormal Results of Clinical Chemistry On Day 3 After Initial Vaccination Compared with Baseline | From initial vaccination up to day 3 post initial vaccination
Percentage of Abnormal Results of Coagulation On Day 3 After Initial Vaccination Compared with Baseline | From initial vaccination up to day 3 post initial vaccination
Percentage of Participants With Any AEs Leading to Discontinuation of Vaccination or Withdrawal From The Study | Through study completion, about 2 years at most

SECONDARY OUTCOMES:
Geometric mean concentration (GMC) for Pre-F Specific IgG Antibody Against RSV A and RSV B | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged ≥60 years)
Geometric Mean Fold Rise (GMFR) for Pre-F Specific IgG Antibody Against RSV A and RSV B | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged ≥60 years)
Seroconversion Rate (SCR) for Pre-F Specific IgG Antibody Against RSV A and RSV B | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged ≥60 years)
Geometric mean titer (GMT) for Neutralizing Antibody Against RSV A and RSV B | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged ≥60 years)
GMFR for Neutralizing Antibody Against RSV A and RSV B | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged ≥60 years)
SCR for Neutralizing Antibody Against RSV A and RSV B | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged ≥60 years)
Frequency of antigen Specific IFN-γ/IL-4 Secreting T cells (Via Enzyme-Linked Immunospot [ELISpot] Assay) | Before vaccination, and 2 weeks and 1, 3 and 6 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3 and 6 months post-initial vaccination (Part 2, participants aged ≥60 years)
Frequency of antigen Specific CD4 and CD8 T Cells Expressing Activation Markers (Via Intracellular Cytokine Staining [ICS] Assay) | Before vaccination, and 2 weeks post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1 month post-initial vaccination (Part 2, participants aged ≥60 years)
Percentage of Participants (Part 2, Aged ≥60 Years) With Solicited Local and Systemic Adverse Reactions Through 14 Days After Revaccination | From second vaccination up to 14 days post revaccination
Percentage of Participants (Part 2, Aged ≥60 Years) With Unsolicited AEs Through 28 Days After Revaccination | From second vaccination up to 28 days post revaccination
Percentage of Participants With AEs Through 30 Minutes After Revaccination (Part 2, Aged ≥60 Years) | From second vaccination up to 30 Minutes post revaccination
Percentage of Abnormal Results of Hematology On Day 3 After Revaccination Compared with Baseline of Revaccination (Part 2, Aged ≥60 Years) | From second vaccination up to Day 3 post revaccination
Percentage of Abnormal Results of Clinical Chemistry On Day 3 After Revaccination Compared with Baseline of Revaccination (Part 2, Aged ≥60 Years) | From second vaccination up to Day 3 post revaccination
Percentage of Abnormal Results of Coagulation On Day 3 After Revaccination Compared with Baseline of Revaccination (Part 2, Aged ≥60 Years) | From second vaccination up to Day 3 post revaccination

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Anning First People's Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided